CLINICAL TRIAL: NCT06035640
Title: Improving Shared Decision Making on the Neonatal Unit Through Assessment of Parental Experiences (The ShAPE Study)
Brief Title: Improving Shared Decision Making on the Neonatal Unit Through Assessment of Parental Experiences
Acronym: ShAPE
Status: Recruiting | Type: Observational
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022/CTU2/NEONAT
Record Dates: First submitted 2023-02-15; First posted 2023-09-13 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Communication
Keywords: Neonatal Care; Shared Decision Making
MeSH Terms: conditions — Communication | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Participants will be engaged in a semi-structured interview.

SUMMARY:
1 in 7 infants born in the United Kingdom will require treatment on a Neonatal unit to treat conditions, which vary in there level of severity. Treatments and interventions aimed at supporting the unwell neonate have associated risks and the evidence underpinning them can range from limited to substantial. There is a degree of uncertainty in Neonatology, which can be very stressful for parents and clinicians alike. Parents need to be supported by the clinical team in making many complicated clinical decisions, a skill that requires robust communication of risks, benefits and alternatives.

In 2019 the British Association of Perinatal Medicine released a framework of care advocating Shared Decision Making (SDM) as the optimal process for making clinical decisions on neonatal units. This model builds upon the "informed decision" models by putting a greater emphasis on involving parents in key decisions regarding the treatment of their babies medical condition. Evidence has demonstrated that SDM can improve parental satisfaction and reduce anxiety and the likelihood of feeling regret.

In order to support parents in the SDM process, clinicians need to be able to provide impartial information encompassing the proposed intervention, intended benefit, potential risks and alternatives. Whilst clinicians may have preconceptions on the information that they think should be provided, there is limited evidence in the literature of what are the most important concepts and themes that parents would expect to be conveyed during the SDM process.

ShAPE is a qualitative study that aims to

ELIGIBILITY:
Inclusion Criteria:

* Parent of an Infant who, whilst on a neonatal unit, has received either; a transfusion of blood products, pharmacotherapy for persistent ductus arteriosus or corticosteroid therapy for chronic lung disease

Exclusion Criteria:

* The infant must have received the above treatments within the last 6 months prior to interview AND have been discharged from neonatal care for at least 4 weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit parents of infants who have received care on a Neonatal Unit within the past 2years. Given the nature of interventions being studied, these are most likely to be (but not limited to) premature infants.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
What are the main communicative, environmental and informative factors that support the facilitation of effective shared decision making on the neonatal unit? We aim to identify common themes that highlight aspects of the decision making process. | Interviews will focus on encounters with clinical staff, whilst their infant was an inpatient on a Neonatal Unit. Interviews will be performed over the 1year period of the recruitment window.
  We aim to identify common themes that highlight aspects of the decision making process, which are the most important to parents.

SECONDARY OUTCOMES:
How does the quality of the shared decision process, experienced by parents on neonatal units in the UK, impact their level of satisfaction with the care their infant received? | Interviews will focus on encounters with clinical staff, whilst their infant was an inpatient on a Neonatal Unit. Interviews will be performed over the 1year period of the recruitment window.
  We aim to identify common themes that highlight aspects of the decision making process, which influence parent satisfaction with the care received by their infant.

CONTACTS AND LOCATIONS:
Locations (1):
- William Harvey Hospital, Ashford, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No